CLINICAL TRIAL: NCT05426330
Title: Cross-sectional, Observational Study of Advanced Cancer Patients' and Their Primary Caregivers' Willingness to Communicate About Advance Care Planning (ACP)
Brief Title: Advanced Cancer Patients' and Their Primary Caregivers' Willingness to Communicate About Advance Care Planning (ACP)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jules Bordet Institute (Other)
Collaborators: Fonds Gaston Ithier (Unknown); Université Libre de Bruxelles (Other); Association Jules Bordet (Unknown)
Responsible Party: Sponsor
Other Study IDs: CE3353
Record Dates: First submitted 2022-05-04; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-04

CONDITIONS: Advanced Cancer
Keywords: Cancer; Advanced Cancer Patients; Primary Caregivers; Advanced Care Planning; ACP; Communication
MeSH Terms: conditions — Neoplasms; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Advanced care planning (ACP) is a major component of end-of-life care. Advanced care planning aims to (1) establish treatment and care options in the event that continuing cancer treatment is more risky than beneficial (e.g., participating in a clinical trial testing a new treatment; continuing supportive care only) and (2) establish possible treatment limitations in the event that a medical complication threatens the patient's survival without the patient's expressed wishes (e.g., transfer to an intensive care unit; resuscitation). However, cancer patients still rarely engage with their physician(s) and family in a discussion about ACP. The primary objective of the project is to conduct a cross-sectional, observational study of the willingness of advanced cancer patients and their primary caregivers to communicate about ACP with each other and with the physician(s); and their agreement/disagreement with these respective willingness. The secondary objective of the project is to assess the medical, psychological and relational factors associated with these willingness. This study will involve 300 consecutive patient- primary caregiver-physician(s) triads. For each patient and their primary caregiver, an in-depth assessment of their willingness to communicate about ACP with each other and with the physician(s) will be conducted using specific scales. The medical, psychological and relational characteristics of the included patients and their primary caregiver will also be assessed using validated questionnaires. Results of this study will enable to propose innovative interventions likely to optimize the establishment of an ACP for numerous advanced cancer patients.

DETAILED DESCRIPTION:
Advanced care planning (ACP) is a major component of end-of-life care. Advanced care planning aims to (1) establish treatment and care options in the event that continuing cancer treatment is more risky than beneficial (e.g., participating in a clinical trial testing a new treatment; continuing supportive care only) and (2) establish possible treatment limitations in the event that a medical complication threatens the patient's survival without the patient's expressed wishes (e.g., transfer to an intensive care unit; resuscitation). ACP aims to ensure that the patient receives care consistent with their personal values, life goals, and preferences. Nowadays, ACP is conceived as an iterative process of communication between patients, their families, and caregivers. However, cancer patients still rarely engage with their physician(s) and family in a discussion about ACP.

There is a gap between the recommendations that communication take place between patients, their families and physician(s) regarding end-of-life care planning, and the application of this recommendation in clinical practice. This gap threatens the quality of life care as well as the adjustment of their caregivers to this phase of the disease and the grief that follows. A thorough and rigorous study of the reasons for this discrepancy has become an essential issue for the oncology of tomorrow.

No studies have quantified the respective willingness of cancer patients and their primary caregivers to communicate about ACP with each other and with their physician(s). No studies have quantified the agreement/disagreement of these patients and their primary caregivers on this issue. No study has assessed the medical, psychological, and relational factors associated with these respective willingness and agreements/disagreements.

This is a cross-sectional observational study. On a weekly basis, the list of eligible patients having a consultation at the Institut Jules Bordet in the medical oncology, hematology, surgery or radiotherapy departments will be provided by the Institute's IT department. An audit of the patients' medical records will be performed by the evaluator. This check will ensure that the patient meets the study's eligibility criteria.

Each patient will be personally contacted by telephone by an evaluator to introduce the study and solicit their participation. During this contact, the patient will identify and provide, if desired, the contact information for their primary caregiver and the physician they designate as their primary decision-maker in the treatment and care of their cancer condition.

A psycho-oncologist evaluator will conduct the assessment for all the patients, their primary caregiver and their physician. This assessment is based on an integrative model of medical, psychological and relational factors associated with the willingness of patients and their relatives to communicate about the patient's ACP. This model has allowed the development of case report forms with different questionnaires. Informed consent forms will be provided by the evaluator, due to the sensitivity of the topics addressed. The questionnaires of the patient, their primary caregiver and their physician will be administered within one month of the first contact with the patient. A simultaneous evaluation will be conducted with patients and primary caregivers. The time difference between the questionnaires of the three protagonists involved in the study will not exceed 72 hours. The completion of the questionnaire will be assisted, in person or if necessary remotely, before the consultation. The survey will be administered using the REDCAP software.

The recruitment of patients, their primary caregiver and their physician will be done consecutively. This recruitment will continue until 300 patient - primary caregiver - physician triads are included in the study. The socio-demographic and medical information of the subjects for whom this evaluation could not be performed, as well as the reasons for this non-evaluation, will be recorded and archived in the study results.

This is the first study to address in a observational manner the willingness of the patient and their primary caregiver to communicate about ACP, their agreement/disagreement with these respective willingness, and the associated medical and relational psychological factors. The Institut Jules Bordet provides a framework for conducting a study, the results of which will allow optimization of the process of establishing an ACP. This optimization will improve the quality of life of these patients and their families. Conducting this study will provide suggestions for interventions that may optimize the establishment of a ACP for many cancer patients.

ELIGIBILITY:
The general eligibility criteria for patients are as follows:

* Be competent (defined according to Appelbaum et al. (1988) as the ability to understand, reason and communicate)
* Speak French
* Be over 18 years of age
* Have given written informed consent to participate in the study

In addition to these general criteria, specific eligibility criteria are defined for patients referred for medical oncology, hematology, surgery or radiotherapy.

Specific criteria for patients attending a medical oncology consultation:

* To have metastatic cancer or cancer with locoregional extension
* and be involved in a new line of treatment (ongoing or planned), following resistance of the disease to at least one first treatment;
* and/or have been diagnosed with brain metastasis.

Specific criteria for patients attending a hematology oncology consultation:

* To have a hemato-oncological condition
* and be involved in a first line of non-curative therapy (e.g. myeloma, acute myeloid leukemia on Vidaza-Venetoclax);
* and/or be involved in a new line of treatment (ongoing or planned), following a relapse of the disease after at least one first line of treatment.

Specific criteria for patients attending a surgery consultation:

* To have metastatic cancer or cancer with locoregional extension
* and be involved in the scheduling of a major surgery.

Specific criteria for patients attending a radiation therapy consultation:

* To have metastatic cancer or cancer with locoregional extension
* and be involved in a radiotherapy treatment involving more than one session

Exclusion Criteria for patients :

* Not being competent (defined according to Appelbaum et al. (1988) as the ability to understand, reason and communicate)
* Have a poor command of the French language
* Already have a therapeutic limitation status, limited to supportive care (BSC status).

Inclusion Criteria for primary Caregivers :

The eligibility criteria for primary caregivers are as follows:

* Have been identified by the patient as the person who supports them the most with their cancer condition
* Be competent
* Speak French
* Be over 18 years of age
* Have given written informed consent to participate in the study

Inclusion Criteria for physicians :

* Have been designated by the patient as the physician with whom they wish to make major decisions in terms of treatment planning and/or therapeutic limitations
* Speak French
* Have given written informed consent to participate in the study

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with advanced cancer who have a consultation at the Institut Jules Bordet in the medical oncology, hematology, surgery or radiotherapy departments.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-10-04 (Estimated); Study Completion 2024-10-04 (Estimated)

PRIMARY OUTCOMES:
Rate of willingness of patients and their primary caregiver to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Willingness to communicate about patients' ACP is assessed through a self-reported questionnaire created for the study and completed by the patients and their primary caregiver named "Willingness to communicate about the patient's ACP". The questionnaire is composed of 8 items regarding the willingness to communicate with each other and with the physician(s) about patients' planification of treatments, care, and the patient's prognosis. Each item has a 4 points Likert scale, ranging from "no" to "yes".
Rate of patients and their primary caregiver's advanced care wishes. | Baseline
  Advanced care wishes are assessed through a self-reported questionnaire created for the study and completed by the patients and their primary caregiver named "advanced care wishes". The questionnaire is composed of 12 items regarding advanced care preferences: participating in a clinical trial, receiving supportive care only, being resuscitated, being transferred to an intensive care unit. Each item has a 4 points Likert scale ranging from "no" to "yes".
Rate of patients and their primary caregiver's perceived self-efficacy to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Perceived self-efficacy to communicate about the patient's ACP is assessed through a self-reported questionnaire created for the study and completed by the patients and their primary caregiver named "Perceived self-efficacy to communicate about the patient's ACP ". The questionnaire is composed of 4 items regarding the patient's and primary caregiver's perception of their efficacy to communicate with each other and with the physician(s) about patient's planification of treatments and care. Each item has a 4 points Likert scale ranging from "no" to "yes".
Rate of patients and their primary caregiver's barriers that prevent them from communicating with each other and with the physician(s) about the patient's ACP. | Baseline
  Barriers that prevent from communicating about the patient's ACP are assessed through a self-reported questionnaire created for the study and completed by the patients and their primary caregiver named "Barriers that prevent from communicating about the patient's ACP". The questionnaire is composed of 14 items regarding the potential barriers that prevent the patients and their primary caregiver from communicating with each other and with the physician(s) about the patient's planification of treatments and care: physical and/or psychological health, religious and/or philosophical beliefs, lack of time and/or availability of the physician(s). Each item has a 4 points Likert scale ranging from "no" to "yes".

SECONDARY OUTCOMES:
Impact of patients and their primary caregiver's socio-demographic characteristics on their willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Socio-demographic characteristics are assessed through a self-reported questionnaire created for the study and completed by the patient and the primary caregiver named "Socio-demographic characteristics". The questionnaire is composed of 14 to 20 items depending on the branching logic: age, gender, current language, cultural background, education and occupation, family status, current and/or previous role as primary or secondary caregiver in the context of a critical illness, previous or ongoing psychological and/or psychiatric support, prior completion of an advanced declaration for euthanasia and identification of a proxy.
Impact of the physician's socio-professional characteristics on patients' and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Socio-professional characteristics are assessed through a self-reported questionnaire created for the study and completed by the physician named "Socio-professional characteristics". The questionnaire is composed of 9 to 11 items depending on the branching logic: age, gender, family status, occupation, clinical practice with advanced cancer patients, professional experience and training, prior completion of an advanced declaration of euthanasia.
Impact of patient's current functional status on patients and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Patients' current functional status is assessed wit the Palliative Performance Scale, composed of 11 items. The scale ranges from "100%" to "0%". A higher score reflects full ambulation, normal activity & work, no evidence of disease, full self-care, normal intake, full conscious level.
Impact of medical factors on patients and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Medical factors are extracted from the patient's chart by the investigator and reported on a specific questionnaire named "Medical characteristics". The questionnaire is composed of 29 items regarding medical history, diagnosis, stage of disease, previous and ongoing cancer treatments.
Impact of perception of the patient's medical situation on patients and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Perception of the patient's medical situation is assessed through a validated self-reported questionnaire adapted for the study and completed by the patients, their primary caregiver and physician(s) named "perception of the patient's medical situation". The questionnaire is composed of 2 to 10 items depending on the branching logic, assess the knowledge about a possibility of cure for the patient's cancer, as well as an estimation of the patient's prognosis.
Impact of physician's communication about the patient's ACP on patients and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Physician's communication about the patient's ACP is assessed through a self-reported questionnaire created for the study and completed by physicians named "Willingness to communicate about the patient's ACP". The questionnaire is composed of 2 items regarding the willingness to communicate with the patient's about his/her planification of care, and about his/her prognosis. Each item has a 4 points Likert scale, ranging from "no" to "yes".
Impact of emotional distress on patients and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Patient's and primary caregiver's emotional distress is assessed with the Hospital Anxiety and Depression Scale (HADS), a 14 items questionnaire, composed by two dimensions (anxiety and depression) and has a 4 point Likert scale that vary at each item. HADS provides a total score (0-42 range) by summing all item scores. A higher score reflects a higher emotional distress. Anxiety subscale score (0-21 range) is provided by summing all Anxiety-items. A higher score reflects more anxiety. Depression subscale scores (0-21 range) is provided by summing all Depression-items. A higher score reflects more depression.
Impact of satisfaction with cancer care on patients and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Satisfaction with cancer care is assessed through a single item from the self-reported questionnaire EORTC QLQ-C-30 and a specific satisfaction questionnaire composed with 10 items and created for the study and completed by the patients and their primary caregiver. Each item has a 5 points Likert scale, ranging from "low" to "excellent".
Impact of Intolerance of Uncertainty on patients and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Intolerance of Uncertainty is assessed through with the Intolerance of Uncertainty Scale - Short Form completed by patients, their primary caregivers, and physicians. This validated questionnaire is composed of 11 items. Each item has a 5 points Likert scale, ranging from "Not at all characteristic of me" to "Entirely characteristic of me".
Impact of moral principles on patients and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Moral principles are assessed through a specific questionnaire of moral dilemma created for the study and completed by patients, their primary caregivers, and physicians. The questionnaire is composed of 4 items corresponding to four hypothetical situations of treatment choice, in which a choice has to be made between two courses of action, either of which entails transgressing the moral principle of autonomy. These situations are written with varying levels of uncertainty. Each item has 2 options: I accept or refuse the treatment.
Impact of decision-making preferences regarding medical decisions on patients and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Decision-making preferences regarding medical decisions are assessed through a validated self-reported questionnaire, the"Control Preference Scale" and completed by patients, their primary caregivers, and physicians. The questionnaire is composed of 2 items regarding who should make decisions regarding the patient's treatment or care (1) if his treatments are more harmful than beneficial, or (2) if in this context a life-threatening medical complication occurs, and the patient cannot express his wishes. Each item has a 7 points Likert scale, ranging from "decisions must be made by myself" to "decisions must be made by myself with my primary caregiver and my physician".
Impact of physicians' perceived self-efficacy to communicate about the patient's ACP on patients and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Perceived self-efficacy to communicate about the patient's ACP is assessed through a self-reported visual analog scale created for the study and completed by physicians named "Perceived self-efficacy to communicate about the patient's ACP". The questionnaire is composed of 3 Visual Analogic Scale (VAS) regarding the physicians' perception of their efficacy to communicate with the patients about their planification of treatments, care, and prognostic. Each VAS ranges from "not at all" to "completely".
Impact of physicians' perceived communication about patients' ACP on patients and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Perceived communication about patients' ACP is assessed through a self-reported visual analog scales (VAS) questionnaire created for the study and completed by physicians named "Perceived communication about patients' ACP". The questionnaire is composed of 3 VAS regarding the stress that the physician may experience when communicating with cancer patients about their advanced care planning and prognostic. Each visual analog scale ranges from "not stressful at all" to "extremely stressful".
Impact of physicians' outcome expectancies regarding communication about patients' ACP on patients and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Perceived outcome expectancies regarding communication about patients' ACP is assessed through a self-reported questionnaire created for the study and completed by physicians named "Perceived communication about patients' ACP". The questionnaire is composed of 12 items regarding the probability of occurrence of specific consequences of the communication with patients about their advanced care planning and prognostic. These consequences are: helping the patients, compromising their coping with cancer, obtaining useful information, or feeling responsible for solving all the concerns expressed. Each has a 5 points Likert scale, ranging from "unlikely" to "very likely".
Impact of collusion between patient, their primary caregiver and the physician(s) on patient, their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Collusion between patient and their caregiver is assessed through a specific questionnaire created for the study and completed by patients and their primary caregivers named "Collusion between patient and their caregiver". The questionnaire is composed of 2 items regarding the respective patient's and caregiver's willingness that the other communicate with the physician(s) about patient's planification of treatments and care. Each item has a 4 points Likert scale ranging from "no" to "yes".
Impact of physician cognitive empathy on patients and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Physician cognitive empathy is assessed through a specific questionnaire created for the study and completed by physicians named "physician's perception of patient's treatment choices". The questionnaire is composed of 1 item regarding the treatment choice the physician would make if he/she was currently in the patient's situation. This item has a 2 options: continuing treatments versus receiving supportive care only.
Impact of physicians' burn out on patients and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Physicians' burn out is assessed with the Maslach Burn Out Inventory (MBI). This validated inventory has three subscales: emotional exhaustion (9 items), depersonalization (5 items) and personal achievement (8 items). Each scale measures its own unique dimension of burnout, using 7 level frequency ratings from "never" to "daily". MBI provides a score on each dimension. A high score on the first two scales and a low score on the last one indicates burnout.
Impact of relational factors on patients and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP. | Baseline
  Relational factors are assessed through a specific questionnaire created for the study and completed by patients and their primary caregivers named "Relationship between the patient, the primary caregiver, and physician(s)". The questionnaire is composed of 6 items regarding: the relationship between the primary caregiver, the patient and the physicians; the time and frequency with which the caregiver helps the patient cope with cancer-related difficulties; the type of help the patient receives (informative, emotional, practical); the frequency with which the patient discusses cancer-related difficulties with the caregiver; date since the physician(s) took care of the patient; number of consultations between the physician(s) and the patient since the start of care.
Impact of perceived daily burden on patients and their primary caregiver's willingness to communicate with each other and with the physician(s) about the patient's ACP | Baseline
  Perceived daily burden is assessed through a self-reported visual analog scale (VAS) created for the study and completed by patients and their primary caregivers named "Perceived daily burden". The questionnaire is composed of 2 items regarding the feeling of being a burden and the feeling of having a burden. The visual analog scale ranges from "not at all" to "completely".

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Appelbaum PS, Grisso T. Assessing patients' capacities to consent to treatment. N Engl J Med. 1988 Dec 22;319(25):1635-8. doi: 10.1056/NEJM198812223192504. PMID 3200278
- [Background] Bhatt VR. Understanding patients' values and priorities in selecting cancer treatments: Developing a therapy preference scale. J Geriatr Oncol. 2019 Sep;10(5):677-679. doi: 10.1016/j.jgo.2018.11.005. Epub 2018 Nov 27. No abstract available. PMID 30501985
- [Background] Bredart A, Beaudeau A, Young T, Moura De Alberquerque Melo H, Arraras JI, Friend L, Schmidt H, Tomaszewski KA, Bergenmar M, Anota A, Costantini A, Marchal F, Tomaszewska IM, Vassiliou V, Chie WC, Hureaux J, Conroy T, Ramage J, Bonnetain F, Kulis D, Aaronson NK; EORTC Quality of Life Group. The European organization for research and treatment of cancer - satisfaction with cancer care questionnaire: revision and extended application development. Psychooncology. 2017 Mar;26(3):400-404. doi: 10.1002/pon.4127. Epub 2016 Apr 13. No abstract available. PMID 27546090
- [Background] Christensen JF, Flexas A, Calabrese M, Gut NK, Gomila A. Moral judgment reloaded: a moral dilemma validation study. Front Psychol. 2014 Jul 1;5:607. doi: 10.3389/fpsyg.2014.00607. eCollection 2014. PMID 25071621
- [Background] Colquitt JA, LePine JA, Noe RA. Toward an integrative theory of training motivation: a meta-analytic path analysis of 20 years of research. J Appl Psychol. 2000 Oct;85(5):678-707. doi: 10.1037/0021-9010.85.5.678. PMID 11055143
- [Background] Degner LF, Sloan JA, Venkatesh P. The Control Preferences Scale. Can J Nurs Res. 1997 Fall;29(3):21-43. PMID 9505581
- [Background] Epstein RM, Duberstein PR, Fenton JJ, Fiscella K, Hoerger M, Tancredi DJ, Xing G, Gramling R, Mohile S, Franks P, Kaesberg P, Plumb S, Cipri CS, Street RL Jr, Shields CG, Back AL, Butow P, Walczak A, Tattersall M, Venuti A, Sullivan P, Robinson M, Hoh B, Lewis L, Kravitz RL. Effect of a Patient-Centered Communication Intervention on Oncologist-Patient Communication, Quality of Life, and Health Care Utilization in Advanced Cancer: The VOICE Randomized Clinical Trial. JAMA Oncol. 2017 Jan 1;3(1):92-100. doi: 10.1001/jamaoncol.2016.4373. PMID 27612178
- [Background] Finkelstein EA, Baid D, Cheung YB, Schweitzer ME, Malhotra C, Volpp K, Kanesvaran R, Lee LH, Dent RA, Ng Chau Hsien M, Bin Harunal Rashid MF, Somasundaram N. Hope, bias and survival expectations of advanced cancer patients: A cross-sectional study. Psychooncology. 2021 May;30(5):780-788. doi: 10.1002/pon.5675. Epub 2021 Apr 1. PMID 33739561
- [Background] Freeston, M. H., Rhéaume, J., Letarte, H., Dugas, M. J., & Ladouceur, R. (1994). Why do people worry? Personality and Individual Differences, 17(6), 791-802. https://doi.org/10.1016/0191-8869(94)90048-5
- [Background] Fried TR, O'Leary JR. Using the experiences of bereaved caregivers to inform patient- and caregiver-centered advance care planning. J Gen Intern Med. 2008 Oct;23(10):1602-7. doi: 10.1007/s11606-008-0748-0. Epub 2008 Jul 30. PMID 18665427
- [Background] Pautex S, Vayne-Bossert P, Bernard M, Beauverd M, Cantin B, Mazzocato C, Thollet C, Bollondi-Pauly C, Ducloux D, Herrmann F, Escher M. Validation of the French Version of the Edmonton Symptom Assessment System. J Pain Symptom Manage. 2017 Nov;54(5):721-726.e1. doi: 10.1016/j.jpainsymman.2017.07.032. Epub 2017 Jul 25. PMID 28751077
- [Background] Razavi, D., Delvaux, N., Farvacques, C., & Robaye, E. (1989). Validation de la version française du HADS dans une population de patients cancéreux hospitalisés [Validation of the French version of the Hospital Anxiety and Depression Scale (HADS) in a population of hospitalized cancer patients]. Revue de Psychologie Appliquée, 39(4), 295-307.
- [Background] Rose JH, O'Toole EE, Dawson NV, Lawrence R, Gurley D, Thomas C, Hamel MB, Cohen HJ. Perspectives, preferences, care practices, and outcomes among older and middle-aged patients with late-stage cancer. J Clin Oncol. 2004 Dec 15;22(24):4907-17. doi: 10.1200/JCO.2004.06.050. Epub 2004 Nov 1. PMID 15520054
- [Background] Sudore RL, Lum HD, You JJ, Hanson LC, Meier DE, Pantilat SZ, Matlock DD, Rietjens JAC, Korfage IJ, Ritchie CS, Kutner JS, Teno JM, Thomas J, McMahan RD, Heyland DK. Defining Advance Care Planning for Adults: A Consensus Definition From a Multidisciplinary Delphi Panel. J Pain Symptom Manage. 2017 May;53(5):821-832.e1. doi: 10.1016/j.jpainsymman.2016.12.331. Epub 2017 Jan 3. PMID 28062339
- [Background] Temel JS, Greer JA, Admane S, Solis J, Cashavelly BJ, Doherty S, Heist R, Pirl WF. Code status documentation in the outpatient electronic medical records of patients with metastatic cancer. J Gen Intern Med. 2010 Feb;25(2):150-3. doi: 10.1007/s11606-009-1161-z. Epub 2009 Nov 6. PMID 19894078
- [Background] Yennurajalingam S, Rodrigues LF, Shamieh OM, Tricou C, Filbet M, Naing K, Ramaswamy A, Perez-Cruz PE, Bautista MJS, Bunge S, Muckaden MA, Fakrooden S, Sewram V, Tejedor AN, Rao SS, Williams JL, Liu DD, Park M, Lu Z, Cantu H, Hui D, Reddy SK, Bruera E. Decisional control preferences among patients with advanced cancer: An international multicenter cross-sectional survey. Palliat Med. 2018 Apr;32(4):870-880. doi: 10.1177/0269216317747442. Epub 2017 Dec 13. PMID 29235415